CLINICAL TRIAL: NCT05508074
Title: A Double-blind, Placebo-controlled, Exploratory Randomised Clinical Trial to Assess the Safety and Efficacy of IFB-088 Plus Riluzole 100 mg vs Placebo Plus Riluzole 100 mg in Patients With Bulbar-onset Amyotrophic Lateral Sclerosis.
Brief Title: Treatment Combining Riluzole and IFB-088 in Bulbar Amyotrophic Lateral Sclerosis (TRIALS Protocol)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InFlectis BioScience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P288ALS; 2021-003875-32 (EudraCT Number)
Record Dates: First submitted 2022-07-27; First posted 2022-08-19 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: IFB-088; Icerguastat; ALS; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neurodegenerative Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neurodegenerative Diseases | interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 2:1 allocation ratio to receive either IFB-088 + riluzole 100 mg or placebo + riluzole 100 mg.
Who Masked: Participant, Investigator
Masking Description: Study double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IFB-088 50 mg/day + riluzole 100 mg/day (Experimental): The test product, IFB-088, will be administered orally in 50 mg/day dosage consisting of two uptakes of 25 mg each (morning and evening uptakes), as an add-on therapy to riluzole 100 mg.
  Intervals for dosing should ideally be about 12 hours (± one hour). Tablets will be swallowed with a glass of water 30 minutes before the meal, in fasting condition.
  Administration of riluzole 100 mg, tablet or suspension, will be at the patient's and/or investigator's choice, as per summary of product characteristics. The daily dose of 100 mg will be taken in two 50 mg doses every 12 hours, at the same time than the IMPs.
  Patients will be treated for a period of 6 months (26 weeks).
  Interventions: Drug: IFB-088 50mg/day; Drug: Riluzole 100mg/day
- placebo + riluzole 100 mg/day (Placebo Comparator): The placebo will be administered orally in two uptakes (morning and evening uptakes), as an add-on therapy to riluzole 100 mg.
  Intervals for dosing should ideally be about 12 hours (± one hour). Tablets will be swallowed with a glass of water 30 minutes before the meal, in fasting condition.
  Administration of riluzole 100 mg, tablet or suspension, will be at the patient's and/or investigator's choice, as per summary of product characteristics. The daily dose of 100 mg will be taken in two 50 mg doses every 12 hours, at the same time than the IMPs.
  Patients will be treated for a period of 6 months (26 weeks).
  Interventions: Drug: Placebo; Drug: Riluzole 100mg/day

INTERVENTIONS:
Drug: IFB-088 50mg/day — Tested product
  Other Names: IFB-088; Icerguastat
  Arms: IFB-088 50 mg/day + riluzole 100 mg/day
Drug: Placebo — Placebo
  Arms: placebo + riluzole 100 mg/day
Drug: Riluzole 100mg/day — Standard of care treatment, co-administered with tested product (IFB-088 50mg/day) or placebo
  Other Names: Riluzole

SUMMARY:
Prospective, international, randomised, double-blind, placebo controlled, multicentre, parallel group study. Patients will be randomised in a 2:1 allocation ratio to receive either IFB-088 + riluzole 100 mg or placebo + riluzole 100 mg. This clinical trial is an exploratory study, designed to show a signal of efficacy of IFB-088 through ALSFRS-R, MITOS and King's College. Respiratory function will be followed through SVC. Biomarkers and quality of life will also be evaluated throughout the study.

Patients will be treated over a 6-month period. After a screening/consent visit, patients will undergo clinic visits at randomisation (V0), at 2 weeks (V1), and at months 1 (V2), 3 (V3) and 6 (V4). One week after V0, the patient will undergo urine analysis (dipstick)and blood sampling for measurement of creatinine

, as well as blood sampling for measurement of creatinine and calculation of eGFR at months 2, 4 and 5. At the V2 visit, in addition to other assessments, patients will undergo blood sampling for PK measurements and urine sampling for crystalluria examination. Blood and urine chemistry, as well as physical examination and vital signs assessment to assess safety will be performed at each visit for safety purpose and crystalluria examination will be repeated at the follow-up visit, performed one month ± one week after V4.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable or definite ALS according to the revised El Escorial criteria [29], with bulbar onset of disease, familial or sporadic form,
2. Onset of symptoms ≤ 18 months prior to screening, as reported by the patient,
3. Adult males or females, aged at least 18 years old,
4. SVC > 60% of predicted value for age and sex,
5. ALSFRS-R score ≥ 36,
6. Treatment with riluzole 100 mg/day, at stable dose since at least one month and well tolerated,
7. Male or female patient of childbearing potential10 who agrees to use highly effective mechanical contraception methods (sexual abstinence, intrauterine device, bilateral tubal occlusion, vasectomised partner) throughout the study, and for 3 months after the end of the treatment,
8. Patient who read, understood and signed the ICF,
9. Patient who is willing to adhere to the study visit schedule and is capable to understand and comply with protocol requirements.

Exclusion Criteria:

1. Known other significant neurological disease(s),
2. Serious illness(es) or medical condition(s) (e.g. unstable cardiac disease, cancer, hematologic disease, hepatitis or liver failure, renal failure) that is not stabilised or that could require hospitalisation and may jeopardise the participation in the study,
3. Abnormal renal function at screening defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2,
4. Abnormal liver function at screening defined as total bilirubin levels >1.5 ULN, and/or AST and/or ALT >3 ULN,
5. Neutropenia (ANC <1.5 x 109/L) at screening,
6. Other causes of neuromuscular weakness,
7. Non progressive or very rapidly progressing ALS (ALSFRS-R decline from disease onset to randomisation ≤ 0.1 / month or ≥ 1.2 / month)11,
8. Non-invasive ventilation,
9. Tracheotomy,
10. Weight loss ≥ 10% compared to weight at symptoms onset as declared by the patient or BMI <18 kg/m2 at screening,
11. Dementia or other severe active psychiatric illness, including suicidal ideation assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS),
12. Patient with a significant pulmonary disorder not attributed to ALS or who require treatments that might complicate the evaluation of the effect of ALS on respiratory function,
13. Patient treated by edaravone for ALS,
14. Patient using unauthorised concomitant treatments, namely moderate or strong inhibitors or inducers of CYP1A2, strong inhibitors or inducers of CYP2D6 or 2C19 and strong inhibitors of OCT2, as listed in Section 6.2. Combined oral contraceptives containing ethinylestradiol are forbidden concomitant medications,
15. Smoker of > 10 cigarettes per day (e-cigarettes and nicotine patches are permitted),
16. Known hypersensitivity to any of the ingredients or excipients of the IMPs,
17. Pregnant, lactating women,
18. Patient who participated in another trial of investigational drug(s) within 30 days prior to randomisation, or 5 half-lives of the previous investigational product, whichever is longer,
19. Patient who has forfeited their freedom by administrative or legal award, or who is under guardianship or under limited judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Attarian, Pr, Principal Investigator — Assistance Publique Hôpitaux de Marseille (APHM) Hospital La Timone Adultes, France; Giuseppe Lauria, Pr, Principal Investigator — IRCCS Carlo Besta Institute of Milan, Italy
Locations (9):
- France (5):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - APHM Hôpital La Timone Adultes SCE Maladies Neuromusculaires / SLA, Marseille
  - CHU de Nantes - Hôpital Laennec, Nantes
  - CHU de Toulouse - Hôpital Pierre-Paul Riquet, Toulouse
  - CHU Bretonneau, Tours
- Italy (4):
  - Ospedale Civile Sant'Agostino Estense, Baggiovara
  - Centro Clinico NeMO per le Malattie Neuromuscolari, Gussago
  - IRCSS Istituto Neurologico Carlo Besta, Milan
  - Sant'Andrea Hospital Unit of Neuromuscular Disorders, Roma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Riluzole 100 mg/Day: The placebo will be administered orally in two uptakes (morning and evening uptakes), as an add-on therapy to riluzole 100 mg.
  Intervals for dosing should ideally be about 12 hours (± one hour). Tablets will be swallowed with a glass of water 30 minutes before the meal, in fasting condition.
  Administration of riluzole 100 mg, tablet or suspension, will be at the patient's and/or investigator's choice, as per summary of product characteristics. The daily dose of 100 mg will be taken in two 50 mg doses every 12 hours, at the same time than the IMPs.
  Patients will be treated for a period of 6 months (26 weeks).
  Placebo: Placebo
  Riluzole 100mg/day: Standard of care treatment, co-administered with tested product (IFB-088 50mg/day) or placebo
- IFB-088 50 mg/Day + Riluzole 100 mg/Day: The test product, IFB-088, will be administered orally in 50 mg/day dosage consisting of two uptakes of 25 mg each (morning and evening uptakes), as an add-on therapy to riluzole 100 mg.
  Intervals for dosing should ideally be about 12 hours (± one hour). Tablets will be swallowed with a glass of water 30 minutes before the meal, in fasting condition.
  Administration of riluzole 100 mg, tablet or suspension, will be at the patient's and/or investigator's choice, as per summary of product characteristics. The daily dose of 100 mg will be taken in two 50 mg doses every 12 hours, at the same time than the IMPs.
  Patients will be treated for a period of 6 months (26 weeks).
  IFB-088 50mg/day: Tested product
  Riluzole 100mg/day: Standard of care treatment, co-administered with tested product (IFB-088 50mg/day) or placebo
Period: Overall Study
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
Started | 17 | 34
Completed | 14 | 23
Not Completed | 3 | 11
Not completed — Death | 2 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — wrongly randomized | 0 | 1
Not completed — non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.6) | 61.1 (11.0) | 62.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 22
  Male | 18 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 17 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 14 | 9 | 23
  France | 20 | 8 | 28
BMI [Median (Standard Deviation); unit: kg/m^2] | 24.49 (3.60) | 23.88 (4.12) | 24.29 (3.75)
Tobacco smoking, n (%) [Count of Participants; unit: Participants]
  Missing data | 0 | 1 | 1
  No | 30 | 16 | 46
  Yes | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessment of IFB-088 50 mg/Day in Patients With Bulbar-onset ALS. Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: * Incidence, grade and relationship to IFB-088 for treatment emergent AEs (TEAEs), SAEs, and AESIs,
  * AEs leading to dose interruption or premature discontinuation.
Time Frame: from beginning of IMP intake up to 30 days after stopping the intake, an average of 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
Number analyzed (Participants) | 17 | 34
Participants
  TEAE | 10 | 25
  TEAE related to study drug | 4 | 13
  Serious TEAE | 4 | 8
  Serious TEAE related to study drug | 0 | 2
  Fatal TEAE | 2 | 5
  Fatal TEAE related to study drug | 0 | 2
  Grade 1 TEAE | 7 | 19
  Grade 2 TEAE | 5 | 11
  Grade > or = 3 TEAE | 3 | 10
  Grade > or = 3 TEAE related to study drug | 0 | 3
  Grade > or = 3 serious TEAE | 2 | 8
  Grade >or = 3 serious TEAE related to study drug | 0 | 2
  TEAE leading to temporary discontinuation of study drug | 1 | 1
  TEAE leading to definitive discontinuation of study drug | 0 | 3

2. Secondary Outcome: Efficacy With Scale : ALSFRS-R (ALS Functional Rating Scale Revised)
Description: ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale Revised) 12 items, clinician rated including 5 choices from normal to disabled.
  Maximal score: 48, minimal score: 0 (death)
Time Frame: Efficacy scale from baseline to V3 (3 months) and V4 (6 months).
Population: The presented data are on the Full Analysis Set (FAS), in which the number of patients changed over time as some patients were lost between baseline and V3 or V4 (death, consent withdrawal, ...).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
Number analyzed (Participants) | 17 | 34
score on a scale
  ALSFRS-R Baseline | 43.9 (2.1) | 42.2 (2.7)
  ALSFRS-R V3 visit (3 months): number analyzed (Participants) | 17 | 31
  ALSFRS-R V3 visit (3 months) | 39.5 (5.9) | 36.0 (8.7)
  ALSFRS-R V4 visit (6 months): number analyzed (Participants) | 17 | 24
  ALSFRS-R V4 visit (6 months) | 34.7 (11.0) | 36.1 (4.4)
Statistical Analysis 1: Comparison: Placebo + Riluzole 100 mg/Day vs IFB-088 50 mg/Day + Riluzole 100 mg/Day; primary analysis results based on estimand 1 (see attached SAP); Test type: Other — the primary endpoint was safety hence the study was not powered to show efficacy. statistical analysis was performed to detect signal of efficacy; p = 0.923, ANCOVA; adjusted on baseline ALSFRS-R and treatment; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-7.27 to 6.60], Standard Error of Mean 3.45
Statistical Analysis 2: Comparison: Placebo + Riluzole 100 mg/Day vs IFB-088 50 mg/Day + Riluzole 100 mg/Day; post hoc analysis adjusted on baseline NfL on top of previous parameters; Test type: Other — FAS post hoc; p = 0.65, ANCOVA — post hoc analysis on the FAS population, adjusted on baseline NfL on top of previous parameters; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-5.1 to 8.2], Standard Error of Mean 3.3

3. Secondary Outcome: Efficacy With Scale : ALS_MITOS (ALS Milano-Torino Staging)
Description: ALS_MITOS (Amyotrophic Lateral Sclerosis Milano-Torino Staging) scale scores the total points of points given in 4 domains (movement, swallowing, communicating, breathing), clinician rated. The ALS8MITOS score is determined by the sum of functional score of 1 for each domain, up to 5, being death. The score may go from 0= no functionnal domain lost, up to 5=death (1 to 4 corresponding to the number of domains lost by the patient).
Time Frame: baseline, V3 (3 months), V4 (6 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
Number analyzed (Participants) | 17 | 34
score on a scale
  Baseline | 0 (0) | 0.1 (0.2)
  V3 visit: number analyzed (Participants) | 17 | 31
  V3 visit | 0.1 (0.3) | 0.4 (0.8)
  V4 visit: number analyzed (Participants) | 17 | 24
  V4 visit | 0.6 (1.2) | 0.3 (0.6)
Statistical Analysis 1: Comparison: Placebo + Riluzole 100 mg/Day vs IFB-088 50 mg/Day + Riluzole 100 mg/Day; primary analysis results based on estimand 1 (see attached SAP); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.398, binomial exact method; Mean Difference (Final Values) = -0.118, 95% CI 2-sided [-0.408 to 0.186]

4. Secondary Outcome: Efficacy With Scale : King's College Scale (ALS Staging Form)
Description: King's college Scale (King's ALS staging form), clinician rated, 8 items. 0=best, 5=death
Time Frame: Efficacy scale from baseline to 3 months and 6 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
Number analyzed (Participants) | 17 | 34
score on a scale
  Baseline | 1.6 (0.8) | 2.1 (0.8)
  V3 visit: number analyzed (Participants) | 17 | 31
  V3 visit | 2.1 (1.2) | 2.7 (0.9)
  V4 visit: number analyzed (Participants) | 17 | 24
  V4 visit | 2.8 (1.4) | 3.0 (1.0)
Statistical Analysis 1: Comparison: Placebo + Riluzole 100 mg/Day vs IFB-088 50 mg/Day + Riluzole 100 mg/Day; calculation based on estimand 1 (see SAP); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.835, binomial exact method; Mean Difference (Final Values) = -0.029, 95% CI 2-sided [-0.326 to 0.271]

5. Secondary Outcome: Efficacy Based on Assessment of Respiratory Function (Slow Vital Capacity [SVC])
Description: Assessment of respiratory function (slow vital capacity [SVC]).
Time Frame: Respiratory function at screening, 3 and 6 months.
Population: The presented data are on the Full Analysis Set (FAS), in which the number of patients changed over time as some patients were lost between baseline and V3 or V4 (death, consent withdrawal, ...). SVC is a respiratory test hence patients suffering from ALS were not always able to perform the test.
Measure: Mean (Standard Deviation); unit: percentage of SVC
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
Number analyzed (Participants) | 17 | 34
percentage of SVC
  Baseline | 88.5 (11.3) | 84.7 (17.8)
  V3 visit: number analyzed (Participants) | 16 | 26
  V3 visit | 74.6 (21.7) | 72.9 (18.4)
  V4 visit: number analyzed (Participants) | 14 | 22
  V4 visit | 67.9 (18.4) | 69.8 (18.3)
Statistical Analysis 1: Comparison: Placebo + Riluzole 100 mg/Day vs IFB-088 50 mg/Day + Riluzole 100 mg/Day; based on estimand 1 (see SAP). change of SVC percentage from baseline to 6 months; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.481, ANCOVA; Mean Difference (Final Values) = 5.31, 95% CI 2-sided [-9.72 to 20.34], Standard Error of Mean 7.47

6. Secondary Outcome: Efficacy Based on Assessment of Respiratory Function (Arterial Blood Gases [ABG]), PaCO2)
Description: Assessment of respiratory function (Arterial Blood Gases [ABG]): description of PaCO2 (mmHg), at screening, 3 and 6 months.
Time Frame: Respiratory function at screening, 3 and 6 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of Mercury
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
millimeters of Mercury
  PaCO2 baseline: number analyzed (Participants) | 32 | 17
  PaCO2 baseline | 37.8 (4.0) | 38.5 (4.5)
  PaCO2 V3 Visit: number analyzed (Participants) | 27 | 15
  PaCO2 V3 Visit | 38.0 (3.9) | 39.5 (4.3)
  PaCO2 V4 visit: number analyzed (Participants) | 24 | 14
  PaCO2 V4 visit | 38.7 (3.7) | 38.0 (5.5)

7. Secondary Outcome: Efficacy Based on Assessment of Body Composition (Exploratory)
Description: change of body composition (% of water, muscle, bone in the body) evaluated by bioelectrical impedance
Time Frame: At baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-01

8. Secondary Outcome: Pharmacokinetic Parameters (Area Under Curve [AUC])
Description: Area Under the Curve (AUC (0-12h)) of IFB-088 and its metabolite IFB-139. As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 ng.h/mL.
Time Frame: PK parameters will be analysed after 4 weeks of treatment. Blood samples were collected at V2 (5 samples/patient: pre-IMP dose, and at one, 2, 4 and 6 hours post dose).
Population: As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 ng.h/mL.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
ng.h/mL
  IFB-088 | 63 (61) | 0 (0)
  IFB-139 (metabolite) | 69 (48.9) | 0 (0)

9. Secondary Outcome: Pharmacokinetic Parameters (Cmax)
Description: Maximum observed plasma concentration (Cmax) of IFB-088 and its metabolite IFB-139.
  As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 ng/mL.
Time Frame: as for outcome 8
Population: As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 ng/mL.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
ng/mL
  IFB-088 | 12 (66.4) | 0 (0)
  IFB-139 (metabolite) | 12 (45.9) | 0 (0)

10. Secondary Outcome: Pharmacokinetic Parameters (Tmax)
Description: Time at which maximum plasma concentration (Cmax) of IFB-088 and its metabolite IFB-139 is measured As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 h
Time Frame: as for outcome 8
Population: As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 h.
Measure: Mean (Inter-Quartile Range); unit: h
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
h
  IFB-088 | 1.0 [1.0 to 4.0] | 0 [0 to 0]
  IFB-139 (metabolite) | 1.0 [1.0 to 4.0] | 0 [0 to 0]

11. Secondary Outcome: Pharmacokinetic Parameters (t1/2)
Description: Terminal or apparent terminal half-life (t1/2) of IFB-088 and its metabolite IFB-139.
  As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 h.
Time Frame: as for outcome 8
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
h
  IFB-088 | 4.62 (40.5) | 0 (0)
  IFB-139 (metabolite) | 7.9 (35.4) | 0 (0)

12. Secondary Outcome: Pharmacokinetic Parameters (Clearance)
Description: IFB-088 Apparent systemic clearance calculation (CL/F) As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 L/h.
Time Frame: as for outcome 8
Population: As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 L/h.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
L/h | 580 (73.0) | 0 (0)

13. Secondary Outcome: Pharmacokinetic Parameters (Vd)
Description: IFB-088 Apparent volume of distribution (Vd). As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 L.
Time Frame: PK parameters will be analysed after 4 weeks of treatment.
Population: As study was double blinded, the analysis was done on all the patients, either receiving IFB-088 or placebo.
  Dosage of IFB-088 in patients under placebo was equal to 0 L.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
L | 3722 (57.9) | 0 (0)

14. Secondary Outcome: Biomarkers (TDP-43)
Description: Change in TDP-43 plasmatic concentration from baseline to 6 months, compared to placebo (concentration in pg/mL, technology Simoa®).
Time Frame: At baseline and 6 months.
Reporting Status: Not Posted, anticipated posting 2026-01

15. Secondary Outcome: Biomarkers (Neurofilament Light Chain)
Description: Change in neurofilament (NfL) light chain plasmatic concentration from baseline to 6 months, compared to placebo (concentration in pg/mL, technology Simoa®).
Time Frame: At baseline and 6 months.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
pg/mL
  Baseline | 86.57 [74.60 to 100.45] | 65.29 [50.73 to 84.02]
  V4 visit: number analyzed (Participants) | 23 | 17
  V4 visit | 92.91 [76.51 to 112.34] | 76.19 [61.95 to 93.70]
Statistical Analysis 1: Comparison: IFB-088 50 mg/Day + Riluzole 100 mg/Day vs Placebo + Riluzole 100 mg/Day; based on available data at V4; Test type: Other; p = 0.609, ANCOVA; adjusted geometric mean ratio = 1.04, 95% CI 2-sided [0.89 to 1.21], Standard Error of Mean 1.08

16. Secondary Outcome: Biomarkers (Inflammation Biomarkers)
Description: Inflammation biomarkers (interleukin [IL]-6, tumour necrosis factor-α [TNFα], interferon γ [IFNγ], IL-1β, IL-8, IL-10, monocyte chemoattractant protein-1 [MCP-1], nerve growth factor [NGF], brain-derived neurotrophic factor [BDNF], vascular endothelial growth factor [VEGF]): (concentration of each biomarker in ng/mL, technology Luminex®)).
Time Frame: All assessed at baseline and V4 visit (6 months). Only GDF15, MCP1, BDNF, and TGFb1 also assessed at V3 visit (3 months)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
ng/mL
  GDF15 baseline | 704.26 [565.60 to 876.93] | 580.31 [437.58 to 769.61]
  GDF15 V3 visit: number analyzed (Participants) | 30 | 17
  GDF15 V3 visit | 711.31 [556.90 to 908.54] | 572.30 [421.00 to 777.98]
  GDF15 V4 visit: number analyzed (Participants) | 23 | 17
  GDF15 V4 visit | 704.90 [541.44 to 917.70] | 580.13 [445.10 to 756.11]
  MCP1 baseline | 168.00 [146.12 to 193.16] | 149.61 [117.08 to 191.17]
  MCP1 V3 visit: number analyzed (Participants) | 30 | 17
  MCP1 V3 visit | 163.47 [137.89 to 193.79] | 131.92 [107.57 to 161.78]
  MCP1 V4 visit: number analyzed (Participants) | 23 | 17
  MCP1 V4 visit | 171.21 [145.78 to 201.06] | 127.53 [100.29 to 162.18]
  BDNF baseline | 2348.36 [1768.30 to 3118.70] | 2717.82 [1687.30 to 4377.72]
  BDNF V3 visit: number analyzed (Participants) | 30 | 17
  BDNF V3 visit | 1892.51 [1364.30 to 2625.23] | 2277.30 [1221.31 to 4246.35]
  BDNF V4 visit: number analyzed (Participants) | 23 | 17
  BDNF V4 visit | 1777.28 [1208.59 to 2613.55] | 2717.49 [1673.06 to 4413.92]
  TGFb1 baseline: number analyzed (Participants) | 33 | 16
  TGFb1 baseline | 30524.88 [24598.01 to 37879.82] | 34174.62 [23139.56 to 50472.23]
  TGFb1 V3 visit: number analyzed (Participants) | 30 | 16
  TGFb1 V3 visit | 25955.30 [20552.48 to 32778.39] | 28333.44 [18658.68 to 43024.70]
  TGFb1 V4 visit: number analyzed (Participants) | 22 | 17
  TGFb1 V4 visit | 20906.55 [15906.89 to 27477.63] | 37702.08 [26739.69 to 53158.68]
  8-OxoDG baseline: number analyzed (Participants) | 26 | 15
  8-OxoDG baseline | 203.01 [173.78 to 237.15] | 175.29 [142.60 to 215.49]
  8-OxoDG V4 visit: number analyzed (Participants) | 24 | 15
  8-OxoDG V4 visit | 220.68 [187.12 to 260.27] | 215.11 [159.73 to 289.69]
  FGF21 baseline | 302.11 [187.86 to 485.85] | 274.81 [144.29 to 523.40]
  FGF21 V4 visit: number analyzed (Participants) | 23 | 17
  FGF21 V4 visit | 230.51 [129.51 to 410.28] | 298.73 [163.68 to 545.22]
  NGFR/p75ECD baseline: number analyzed (Participants) | 26 | 15
  NGFR/p75ECD baseline | 5143.46 [4135.27 to 6397.47] | 4281.16 [2994.38 to 6120.91]
  NGFR/p75ECD V4 visit: number analyzed (Participants) | 24 | 15
  NGFR/p75ECD V4 visit | 6675.13 [5401.43 to 8249.19] | 6108.71 [4569.22 to 8166.90]
  IL-6 baseline | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL-6 V4 visit: number analyzed (Participants) | 23 | 17
  IL-6 V4 visit | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  TNFa baseline | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  TNFa V4 visit: number analyzed (Participants) | 23 | 17
  TNFa V4 visit | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IFNg baseline | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IFNg V4 visit: number analyzed (Participants) | 23 | 17
  IFNg V4 visit | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL1b baseline | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL1b V4 visit: number analyzed (Participants) | 23 | 17
  IL1b V4 visit | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL8 baseline | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL8 V4 visit: number analyzed (Participants) | 23 | 17
  IL8 V4 visit | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL10 baseline | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection
  IL10 V4 visit: number analyzed (Participants) | 23 | 17
  IL10 V4 visit | NA [NA to NA] — below the limit of detection | NA [NA to NA] — below the limit of detection

17. Secondary Outcome: Biomarkers (3-Nitrotyrosine)
Description: 3-Nitrotyrosine (Oxidative stress biomarker): at baseline, 3 and 6 months (concentration in ng/mL, ELISA method).
Time Frame: At baseline, 3 months, and 6 months.
Reporting Status: Not Posted, anticipated posting 2026-01

18. Secondary Outcome: Quality of Life With ALSAQ-40 (ALS Assessment Questionnaire)
Description: Change in ALS assessment questionnaire (ALSAQ-40). ALSAQ-40 (Amyotrophic Lateral Sclerosis Assessment Questionnaire) Quality of Life questionnaire 40 items, patient rated including 5 choices from never to always.
  best=0, worse=100
Time Frame: QoL will be assessed from baseline to 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
score on a scale
  Baseline | 40.7 (20.5) | 39.5 (22.3)
  V4 visit: number analyzed (Participants) | 23 | 16
  V4 visit | 67.1 (31.3) | 61.4 (27.5)

19. Secondary Outcome: Efficacy Based on Assessment of Respiratory Function (Arterial Blood Gases [ABG]), PO2 (mmHg)
Description: Assessment of respiratory function (Arterial Blood Gases [ABG]): description of PO2 (mmHg) at screening, 3 and 6 months.
Time Frame: Respiratory function at screening, 3 and 6 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of Mercury
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
millimeters of Mercury
  PaO2 baseline: number analyzed (Participants) | 32 | 17
  PaO2 baseline | 88.8 (16.8) | 97.5 (25.8)
  PaO2 V3 Visit: number analyzed (Participants) | 27 | 15
  PaO2 V3 Visit | 97.4 (24.5) | 89.1 (14.1)
  PaO2 V4 Visit: number analyzed (Participants) | 24 | 14
  PaO2 V4 Visit | 91.6 (12.6) | 93.3 (27.6)

20. Secondary Outcome: Efficacy Based on Assessment of Respiratory Function (Arterial Blood Gases [ABG]), HCO3 (mEq/L)
Description: Assessment of respiratory function (Arterial Blood Gases [ABG]): description of HCO3 (mEq/L) at screening, 3 and 6 months.
Time Frame: Respiratory function at screening, 3 and 6 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mEq/L (HCO3)
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
mEq/L (HCO3)
  HCO3 baseline: number analyzed (Participants) | 31 | 17
  HCO3 baseline | 24.7 (1.9) | 24.8 (1.9)
  HCO3 V3 visit: number analyzed (Participants) | 27 | 15
  HCO3 V3 visit | 24.8 (2.2) | 24.8 (2.7)
  HCO3 V4 visit: number analyzed (Participants) | 24 | 14
  HCO3 V4 visit | 25.5 (2.6) | 24.6 (3.5)

21. Secondary Outcome: Efficacy Based on Assessment of Respiratory Function (Arterial Blood Gases [ABG]), Oxygen Saturation (%)
Description: Assessment of respiratory function (Arterial Blood Gases [ABG]): description of Oxygen saturation (%) at screening, 3 and 6 months.
Time Frame: Respiratory function at screening, 3 and 6 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % (O2 sat)
Arm/Group | IFB-088 50 mg/Day + Riluzole 100 mg/Day | Placebo + Riluzole 100 mg/Day
Number analyzed (Participants) | 34 | 17
% (O2 sat)
  O2 saturation baseline: number analyzed (Participants) | 32 | 17
  O2 saturation baseline | 96 (2.5) | 96.9 (1.7)
  O2 saturation V3 visit: number analyzed (Participants) | 27 | 15
  O2 saturation V3 visit | 95.2 (6.0) | 96.3 (2.1)
  O2 stauration V4 visit: number analyzed (Participants) | 24 | 14
  O2 stauration V4 visit | 96.7 (1.7) | 96.6 (2.2)

ADVERSE EVENTS:
Time Frame: 7 months, from inclusion to last patient visit, one month after 6 months treatment ending
Arm/Group | Placebo + Riluzole 100 mg/Day | IFB-088 50 mg/Day + Riluzole 100 mg/Day
All-Cause Mortality (participants affected / at risk) | 2/17 | 5/34
Serious Adverse Events (participants affected / at risk) | 4/17 | 8/34
Other Adverse Events (participants affected / at risk) | 10/17 | 25/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Riluzole 100 mg/Day (N=17) | IFB-088 50 mg/Day + Riluzole 100 mg/Day (N=34)
COVID 19 (Infections and infestations) | 1 (4) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (8)
Pneumonia aspiration (Infections and infestations) | 1 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (8)
Pneumonia viral (Infections and infestations) | 1 (4) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (8)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (8)
cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (8)
disease progression (General disorders) | 0 (0) | 1 (8)
hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Riluzole 100 mg/Day (N=17) | IFB-088 50 mg/Day + Riluzole 100 mg/Day (N=34)
Nausea (Gastrointestinal disorders) | 1 (10) | 3 (25)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (25)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (10) | 2 (25)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (25)
dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (25)
Abdominal pain upper (Gastrointestinal disorders) | 1 (10) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (25)
reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (25)
hypertension (Vascular disorders) | 0 (0) | 2 (25)
flank pain (Renal and urinary disorders) | 0 (0) | 1 (25)
pollakiuria (Renal and urinary disorders) | 1 (10) | 0 (0)
anxiety (Psychiatric disorders) | 1 (10) | 0 (0)
depression (Psychiatric disorders) | 1 (10) | 0 (0)
mood altered (Psychiatric disorders) | 1 (10) | 0 (0)
asthenia (General disorders) | 0 (0) | 1 (25)
disease progression (General disorders) | 1 (10) | 0 (0)
pyrexia (General disorders) | 1 (10) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (25)
bradycardia (Cardiac disorders) | 0 (0) | 1 (25)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (25)
cardia-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (25)
exostosis (Musculoskeletal and connective tissue disorders) | 1 (10) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (25)
spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (25)
tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (25)
gastrostomy (Surgical and medical procedures) | 2 (10) | 1 (25)
cataract operation (Surgical and medical procedures) | 1 (10) | 0 (0)
hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (25)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (25)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (25)
erythema (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0)
rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (25)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (25)
fall (Injury, poisoning and procedural complications) | 0 (0) | 8 (25)
clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (25)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 1 (25)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (25)
hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (25)
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (25)
lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (25)
lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (25)
orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (10) | 0 (0)
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (10) | 0 (0)
COVID-19 (Infections and infestations) | 2 (10) | 3 (25)
Oral fungal infection (Infections and infestations) | 2 (10) | 1 (25)
bronchitis (Infections and infestations) | 1 (10) | 1 (25)
urinary tract infection (Infections and infestations) | 1 (10) | 2 (25)
bronchitis fungal (Infections and infestations) | 1 (10) | 0 (0)
cystitis (Infections and infestations) | 0 (0) | 1 (25)
device related sepsis (Infections and infestations) | 0 (0) | 1 (25)
diverticulitis (Infections and infestations) | 0 (0) | 1 (25)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (25)
influenza (Infections and infestations) | 0 (0) | 1 (25)
pneumonia (Infections and infestations) | 0 (0) | 1 (25)
pneumonia aspiration (Infections and infestations) | 1 (10) | 0 (0)
pneumonia viral (Infections and infestations) | 1 (10) | 0 (0)
respiratory tract infection (Infections and infestations) | 0 (0) | 1 (25)
sebaceous gland infection (Infections and infestations) | 0 (0) | 1 (25)

LIMITATIONS AND CAVEATS:
Assessment of Body Composition (Exploratory) could not be assessed properly due to late availability of the devices.

Biomarkers analysis performed by the primary laboratory plant lead to important BLQ data, important CV deviations, requiring cautious interpretation of the results.

Additional biomarker analysis were performed in another lab, and were used for post hoc analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT05508074/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT05508074/SAP_001.pdf